CLINICAL TRIAL: NCT01350687
Title: New Phosphore Binders in Prevention of Pulmonary Hypertension
Brief Title: Pulmonary Hypertension Prevention in Hemodialysis
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: The Baruch Padeh Medical Center, Poriya (Other Government)
Responsible Party: Avi On, Poria Medical Center
Other Study IDs: farid.CTIL
Record Dates: First submitted 2011-05-08; First posted 2011-05-10 (Estimated); Last update posted 2011-05-10 (Estimated); Status verified 2011-04

CONDITIONS: Chronic Kidney Disease
Keywords: Calcium Phosphore; Renagel
MeSH Terms: conditions — Renal Insufficiency, Chronic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Pulmonary hypertension is a new complication described in hemodialysis patients. in the last year these patients were treated by calcium carbonate orally to control serum phosphor. Calcium phosphor deposits in pulmonary artery can explain this phenomena. The investigators want to investigate the new phosphor non calcium containing agents in hemodialysis patients and to measure the pulmonary pressure.

DETAILED DESCRIPTION:
The investigators will measure pulmonary blood pressure before and after treatment with new phosphor binders, non calcium containing.

ELIGIBILITY:
Inclusion Criteria:

* Hemodialysis Patients without fistula

Exclusion Criteria:

* Heart Disease

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 40 patients on hemodialysis treated with Phosphore biders, non-calcium containig.
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2011-06; Primary Completion 2013-06 (Estimated); Study Completion 2014-06 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Farid Nakhoul, Prof., Study Chair — Poria medical Center
Locations (1):
- Poria Medical Center, Tiberias, Israel